CLINICAL TRIAL: NCT03431428
Title: Comparison of Short-term Efficacy and Long-term Prognosis for Reduction Surgery and Radical Resection in Almost-cCR Rectal Cancer Patients: A Case-matched Study
Brief Title: Comparison of Short-term Efficacy and Long-term Prognosis for Reduction Surgery and Radical Resection in Almost-cCR Rectal Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhang Rui (Other)
Responsible Party: Sponsor-Investigator, Zhang Rui, Head of colorectal surgery,clinical professor, Liaoning Cancer Hospital & Institute
Organization: Liaoning Cancer Hospital & Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20171112
Record Dates: First submitted 2018-01-13; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2017-12

CONDITIONS: Almost-cCR; Surgery; Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Transanal Endoscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transanal surgery (Experimental): To ensure the complete cutting edge with no residual tumor, the tumor with corresponding mesorectal excision was removed by the distance edge of 1cm.
  The intestinal wall was sutured to ensure the integrity of the bowel.
  Interventions: Procedure: transanal surgery; Drug: Preoperative chemoradiotherapy
- Miles surgery (Placebo Comparator): According to the total mesorectal excision(TME) principle, complete mesorectum, lymph node and the anus was excised. A sigmoid colostomy was finally performed.
  Interventions: Procedure: Miles surgery; Drug: Preoperative chemoradiotherapy

INTERVENTIONS:
Procedure: transanal surgery — Transanal surgery could Preserve anus to reduce trauma and improve the quality of life
  Arms: transanal surgery
Procedure: Miles surgery — Miles surgery cut off the anus, enlarge the trauma and reduce the quality of life.
  Arms: Miles surgery
Drug: Preoperative chemoradiotherapy — After preoperative radiochemotherapy, two cycles of XELOX were given at the interval of waiting operation.

SUMMARY:
The aim of this study is evaluate the effect of two different surgical treatment on lower rectal cancer after almost clinical complete response(almost-cCR). All almost clinical complete response(almost-cCRs) were entered into two groups randomly. The estimated sample size of the minimal operation group was 221, and 221 in the Mile's group. Three years' progression-free survival(PFS) and overall survival(OS) were compared.

DETAILED DESCRIPTION:
Patients with low rectal cancer were treated with neoadjuvant radiotherapy, and two cycles of XELOX at the interval. All almost-cCRs after neoadjuvant treatment were randomly divided into minimal operation group or Mile's group. All cCRs were treated with "watch and wait". Patients after local recurrence were randomly divided into minimal operation group or Mile's group. If pathological result was pathological staging 3 after neoadjuvant therapy（ypT3） in minimal operation group or local postoperative recurrence occurred, patients need supplement of abdominoperineal resection (APR). With 3 years follow-up，the main research goals are 3 years of progression-free survival(PFS) and overall survival(OS). Secondary endpoints are side effects of chemotherapy, assessment of quality of life, surgical complications, adverse prognostic factors and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Histology is confirmed as rectal adenocarcinoma.
2. 18 to 75 years old.
3. Preoperative staging is lower than clinical stage primary tumor grade 3, regional lymph node grade 1, and metastasis was grade 0（cT3cN1M0）.
4. The anus couldn't be retained after TME.
5. Almost-cCR or cCR recurrence during observation.

Exclusion Criteria:

1. Patients were unable to tolerate the operation.
2. Preoperative stage: T4b or progress during the treatment.
3. HIV infection stage or chronic hepatitis B.
4. Active clinical severe infections.
5. Evil liquid state or decompensation of organ function.
6. Other malignant tumor history in five years.
7. Other primary carcinoma.
8. Unstable condition and incompliance of the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | three years
  The progression-free survival of 3 years
OS | three years
  3 years of overall survival time

SECONDARY OUTCOMES:
carcinoembryonic antigen（CEA） | every 3 months,for 2 years
  The level of carcinoembryonic antigen in blood
carbohydrate antigen 19-9（CA-199） | every 3 months,for 2 years
  The level of carbohydrate antigen 19-9 in blood
International Index of Erectile Function-15 | every 3 months ,for 2 years
  Describe the function of Erectile ,only for male patients
International prostate symptom score | every 3 months ,for 2 years
  Describe the function of prostate,only for male patients
Female sexual function index | every 3 months,for 2 years
  Describe the function of sexual for female patients
Wexner incontinence score | every 3 months,for 2 years
  Describe the degree of Anus incontinence
QOL | every 3 months,for 2 years
  Describe the quality of life for tumor patients

CONTACTS AND LOCATIONS:
Overall Officials: peirong ding, doctor, Principal Investigator — Sun Yat-sen University; ji zhu, doctor, Principal Investigator — Fudan University; zhenning wang, doctor, Principal Investigator — First Hospital of China Medical University; hong zhang, doctor, Principal Investigator — Shengjing Hospital; yu han, doctor, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University; zhaocheng chi, doctor, Principal Investigator — Jilin Provincial Tumor Hospital; quan wang, doctor, Principal Investigator — The First Bethune Hospital of Jilin University; ge liu, doctor, Principal Investigator — The First Affiliated Hospital of Dalian Medical University; hang lu, doctor, Principal Investigator — Jinzhou Medical University; zheng liu, doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; rui Zhang, doctor, Study Director — Liaoning Cancer Hospital & Institute
Locations (1):
- Liaoning cancer Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Motamedi MAK, Mak NT, Brown CJ, Raval MJ, Karimuddin AA, Giustini D, Phang PT. Local versus radical surgery for early rectal cancer with or without neoadjuvant or adjuvant therapy. Cochrane Database Syst Rev. 2023 Jun 13;6(6):CD002198. doi: 10.1002/14651858.CD002198.pub3. PMID 37310167